CLINICAL TRIAL: NCT03011515
Title: A Multi-center, Prospective, Validation Study to Assess the Accuracy of a Host-response Based Diagnostic for Distinguishing Between Bacterial and Viral Etiology in Adult Patients With Lower Respiratory Tract Infections
Brief Title: Evaluating a Host-response Based Diagnostic for Distinguishing Between Bacterial and Viral Etiology in Patients With Lower Respiratory Tract Infection (LRTI)
Acronym: OBSERVER
Status: Completed | Type: Observational
Sponsor: MeMed Diagnostics Ltd. (Industry)
Collaborators: Rambam Health Care Campus (Other); Carmel Medical Center (Other); Rabin Medical Center (Other); European Commission (Other)
Responsible Party: Sponsor
Other Study IDs: MM-1005-OB
Record Dates: First submitted 2017-01-04; First posted 2017-01-05 (Estimated); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Lower Respiratory Tract Infection; Acute Bronchitis; Pneumonia; Chronic Obstructive Pulmonary Disease (COPD); Upper Respiratory Tract Infection
MeSH Terms: conditions — Bronchitis; Pneumonia; Pulmonary Disease, Chronic Obstructive; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood and nasal swab
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- LRTI patients: Patients with suspicion of LRTI, excluding episodes of COPD exacerbations
- Non-infectious patients: Afebrile patients with no apparent infectious disease
- LRTI patients with COPD: Patients with suspicion of LRTI in a sub-group of patients with COPD

SUMMARY:
The purpose of this study is to validate the diagnostic accuracy of a novel host-response based diagnostic tool for differentiating between bacterial and viral etiologies in adult patients aged 18 years and older with clinical suspicion of lower respiratory tract infections (LRTI)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older who agree (or their legal guardian agree) to sign an informed consent will be eligible for inclusion.
* The LRTI cohorts should also fulfill the following criteria:

  * Peak measured (not tactile, self-reported acceptable) temperature ≥ 37.8°C (100°F) within the last 7 days (AND)
  * Symptoms duration ≤7 days (AND)
  * Clinical suspicion of LRTI or pneumonia

Exclusion Criteria:

* Oral/intravenous/intramuscular antibiotic treatment of over 48/12/12 hours' duration at time of enrollment (respectively), unless temperature ≥ 37.8°C was measured within the last 2 days
* Another episode of an acute infection during the last 2 weeks
* Congenital immune deficiency (CID)
* A proven or suspected human immunodeficiency virus (HIV)-1, hepatitis B virus (HBV), or hepatitis C virus (HCV) infection
* Active malignancy
* Pregnancy
* Current treatment with immune-suppressive or immune-modulating therapies including without limitations:

  * Use of high dose steroids >1 mg/kg/day prednisone or equivalent in the past two weeks
  * Monoclonal antibodies
  * Intravenous immunoglobulin (IVIG)
  * Cyclosporine, Cyclophosphamide, Tacrolimus
  * Granulocyte/Monocyte colony stimulating factor (G/GM-CSF)
  * Anti-Tumor Necrosis Factor (TNF) agents
  * Interferon (of all kinds)
* Other severe illnesses that affect life expectancy and quality of life such as:

  * Moderate to severe psychomotor retardation
  * Post-transplant patients (including solid organs, allogeneic/autologous stem cell transplantation)
  * Moderate to severe congenital metabolic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include eligible patients aged 18 years and older of both genders that attend the emergency department or affiliated community clinics due to a suspected LRTI, or due to a non-infectious disease.
Sampling Method: Non-Probability Sample
Enrollment: 583 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
To externally validate the diagnostic accuracy of a host-response based diagnostic tool called ImmunoXpert™, for differentiating between bacterial and viral etiologies in adult patients aged 18 years and older with clinical suspicion of LRTI | 0-6 days after the initiation of symptoms

SECONDARY OUTCOMES:
To compare the diagnostic accuracy of ImmunoXpert™ to currently available lab measures (WBC, ANC, PCT, CRP), using sensitivity and specificity measures and predetermined cutoffs | 0-6 days after the initiation of symptoms
To compare ImmunoXpert™ results with the physician suspected diagnosis at time of patient recruitment and compared to the reference standard diagnosis | 0-6 days after the initiation of symptoms
To estimate the potential improvement in health and economic outcomes following the usage of ImmunoXpert™ compared to current practice | 0-6 days after the initiation of symptoms
To estimate the diagnostic accuracy of ImmunoXpert™ in differentiating between infectious vs non-infectious patients | 0-6 days after the initiation of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Mical Paul, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

REFERENCES:
- [Background] Oved K, Cohen A, Boico O, Navon R, Friedman T, Etshtein L, Kriger O, Bamberger E, Fonar Y, Yacobov R, Wolchinsky R, Denkberg G, Dotan Y, Hochberg A, Reiter Y, Grupper M, Srugo I, Feigin P, Gorfine M, Chistyakov I, Dagan R, Klein A, Potasman I, Eden E. A novel host-proteome signature for distinguishing between acute bacterial and viral infections. PLoS One. 2015 Mar 18;10(3):e0120012. doi: 10.1371/journal.pone.0120012. eCollection 2015. PMID 25785720
- [Background] Eden E, Srugo I, Gottlieb T, Navon R, Boico O, Cohen A, Bamberger E, Klein A, Oved K. Diagnostic accuracy of a TRAIL, IP-10 and CRP combination for discriminating bacterial and viral etiologies at the Emergency Department. J Infect. 2016 Aug;73(2):177-80. doi: 10.1016/j.jinf.2016.05.002. Epub 2016 May 30. No abstract available. PMID 27255416
- [Background] van Houten CB, de Groot JAH, Klein A, Srugo I, Chistyakov I, de Waal W, Meijssen CB, Avis W, Wolfs TFW, Shachor-Meyouhas Y, Stein M, Sanders EAM, Bont LJ. A host-protein based assay to differentiate between bacterial and viral infections in preschool children (OPPORTUNITY): a double-blind, multicentre, validation study. Lancet Infect Dis. 2017 Apr;17(4):431-440. doi: 10.1016/S1473-3099(16)30519-9. Epub 2016 Dec 22. PMID 28012942
- See also: Related Info — http://www.me-med.com/